CLINICAL TRIAL: NCT00207883
Title: Ultrasound Guided Vascular Access: A Prospective Comparison Study
Brief Title: Ultrasound Guided Vascular Access in Pediatric Intensive Care Patients
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Jana Stockwell, MD, Children's Healthcare of Atlanta
Other Study IDs: 04-130
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Critical Illness
Keywords: Vascular Access; Ultrasound; Pediatric; Pediatric intensive care patient
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Landmark: Procedure/Surgery: Use of landmarks for central line placement
- Ultrasound guided: Procedure/Surgery: Use of ultrasound for central line placement

SUMMARY:
The purpose of this study is to see how fast and accurate two different techniques used by physicians to insert catheters in children are. Catheters are tiny tubes which carry fluids, blood and sometimes liquid food into a person's vein. The technique currently used relies on the physical landmarks and using fingers to feel the anatomy in which to place the catheter in the vein or artery. The investigators are changing to a technique where they will use ultrasound at the patient's bedside to help physicians with placing the catheter into the blood vessel. They are comparing the use of these two methods to determine which is faster and requires fewer needle sticks.

DETAILED DESCRIPTION:
In critically ill patients, central venous access is essential for volume resuscitation, administration of medicines (such as vasoactive drugs, antibiotics or chemotherapy), administration of blood products, and hemodynamic monitoring. Placement of central venous catheters (CVC) occurs commonly with over 200,000 CVCs placed in adults and children yearly. At Egleston 222 central venous lines were placed last year and 178 CVCs YTD through October. Obtaining central venous access in critically ill children can be a difficult procedure with many potential complications. These complications can include, but are not limited to, hematoma at the site, hemothorax, pneumothorax, need to change sites, and injury to surrounding structures. The complication rates for CVCs in children is reported anywhere from 2.5% to 22%. All too frequently CVC placement in children is unsuccessful anywhere from 5% of the time to greater than 19%.

Studies in adults have shown ultrasound guided central venous access to decrease the number of attempts required to cannulate the vein. Ultrasound (US) guidance is also able to decrease the time required to cannulate the vessel. A meta analysis of ultrasound guided central venous access in adults concluded that for internal jugular procedures ultrasound guidance was significantly more successful than the landmark technique alone. With the recent focus on patient safety and clinical outcomes the American College of Emergency Physicians published a policy statement included in the guidelines use of US guidance for central venous access in a list of primary applications for ultrasound in the emergency department.

Evidence for US guidance in children is currently found mainly in the anesthesia literature. The 2003 NICE sponsored meta-analysis showed an overall relative risk reduction of 85% for failed placement and 73% for complications of internal jugular placement in pediatric patients in an operating room. Because of small sample sizes (each < 100 patients) and only the internal jugular approach being studied, definitive conclusions regarding other sites are ongoing. Currently there are no prospective studies evaluating the use of ultrasound guided central venous access in children in a pediatric intensive care unit. Also, studies addressing the use of US guided CVC placement in femoral access, the major site used in children, is also lacking.

Our proposal is to prove that US guided CVC will decrease the overall time required to cannulate the vessel by increasing the probability of successful cannulation by the first operator, decreasing the number of skin punctures to obtain access, eliminating the need to change sites for access, and improving the probability of access. Additionally we believe that US guided CVC placement would decrease the likelihood of untoward effects including but not limited to severe hematoma requiring attempts at additional sites, inadvertent puncture of the wrong vessel, or hemothorax/pneumothorax.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the pediatric intensive care unit (PICU) who require vascular access.

Exclusion Criteria:

* Age greater than 18 years.
* Any vascular catheter placed outside of the pediatric intensive care unit at Egleston.
* Any vascular catheter placed by a physician other than a member of the pediatric critical care team.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients admitted to the Pediatric Intensive care Unit (PICU) at Children's Healthcare of Atlanta at Egleston
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jana A Stockwell, MD, Principal Investigator — Children's Healthcare of Atlanta; Curt Froehlich, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sznajder JI, Zveibil FR, Bitterman H, Weiner P, Bursztein S. Central vein catheterization. Failure and complication rates by three percutaneous approaches. Arch Intern Med. 1986 Feb;146(2):259-61. doi: 10.1001/archinte.146.2.259. PMID 3947185
- [Background] Casado-Flores J, Barja J, Martino R, Serrano A, Valdivielso A. Complications of central venous catheterization in critically ill children. Pediatr Crit Care Med. 2001 Jan;2(1):57-62. doi: 10.1097/00130478-200101000-00012. PMID 12797890
- [Background] Stenzel JP, Green TP, Fuhrman BP, Carlson PE, Marchessault RP. Percutaneous femoral venous catheterizations: a prospective study of complications. J Pediatr. 1989 Mar;114(3):411-5. doi: 10.1016/s0022-3476(89)80559-1. PMID 2921683
- [Background] Venkataraman ST, Thompson AE, Orr RA. Femoral vascular catheterization in critically ill infants and children. Clin Pediatr (Phila). 1997 Jun;36(6):311-9. doi: 10.1177/000992289703600601. PMID 9196229
- [Background] Miller AH, Roth BA, Mills TJ, Woody JR, Longmoor CE, Foster B. Ultrasound guidance versus the landmark technique for the placement of central venous catheters in the emergency department. Acad Emerg Med. 2002 Aug;9(8):800-5. doi: 10.1111/j.1553-2712.2002.tb02168.x. PMID 12153885
- [Background] Milling TJ Jr, Rose J, Briggs WM, Birkhahn R, Gaeta TJ, Bove JJ, Melniker LA. Randomized, controlled clinical trial of point-of-care limited ultrasonography assistance of central venous cannulation: the Third Sonography Outcomes Assessment Program (SOAP-3) Trial. Crit Care Med. 2005 Aug;33(8):1764-9. doi: 10.1097/01.ccm.0000171533.92856.e5. PMID 16096454
- [Background] Leung J, Duffy M, Finckh A. Real-time ultrasonographically-guided internal jugular vein catheterization in the emergency department increases success rates and reduces complications: a randomized, prospective study. Ann Emerg Med. 2006 Nov;48(5):540-7. doi: 10.1016/j.annemergmed.2006.01.011. Epub 2006 Feb 21. PMID 17052555
- [Background] Randolph AG, Cook DJ, Gonzales CA, Pribble CG. Ultrasound guidance for placement of central venous catheters: a meta-analysis of the literature. Crit Care Med. 1996 Dec;24(12):2053-8. doi: 10.1097/00003246-199612000-00020. PMID 8968276
- [Background] Keenan SP. Use of ultrasound to place central lines. J Crit Care. 2002 Jun;17(2):126-37. doi: 10.1053/jcrc.2002.34364. PMID 12096376
- [Background] Hind D, Calvert N, McWilliams R, Davidson A, Paisley S, Beverley C, Thomas S. Ultrasonic locating devices for central venous cannulation: meta-analysis. BMJ. 2003 Aug 16;327(7411):361. doi: 10.1136/bmj.327.7411.361. PMID 12919984
- [Background] Shojania KG, Duncan BW, McDonald KM, Wachter RM, Markowitz AJ. Making health care safer: a critical analysis of patient safety practices. Evid Rep Technol Assess (Summ). 2001;(43):i-x, 1-668. PMID 11510252
- [Background] American College of Emergency Physicians.. American College of Emergency Physicians. Use of ultrasound imaging by emergency physicians. Ann Emerg Med. 2001 Oct;38(4):469-70. doi: 10.1067/mem.2001.118487. No abstract available. PMID 11574809
- [Background] Verghese ST, McGill WA, Patel RI, Sell JE, Midgley FM, Ruttimann UE. Ultrasound-guided internal jugular venous cannulation in infants: a prospective comparison with the traditional palpation method. Anesthesiology. 1999 Jul;91(1):71-7. doi: 10.1097/00000542-199907000-00013. PMID 10422930
- [Background] Verghese ST, McGill WA, Patel RI, Sell JE, Midgley FM, Ruttimann UE. Comparison of three techniques for internal jugular vein cannulation in infants. Paediatr Anaesth. 2000;10(5):505-11. doi: 10.1046/j.1460-9592.2000.00554.x. PMID 11012954
- [Background] Leyvi G, Taylor DG, Reith E, Wasnick JD. Utility of ultrasound-guided central venous cannulation in pediatric surgical patients: a clinical series. Paediatr Anaesth. 2005 Nov;15(11):953-8. doi: 10.1111/j.1460-9592.2005.01609.x. PMID 16238556
- [Background] Grebenik CR, Boyce A, Sinclair ME, Evans RD, Mason DG, Martin B. NICE guidelines for central venous catheterization in children. Is the evidence base sufficient? Br J Anaesth. 2004 Jun;92(6):827-30. doi: 10.1093/bja/aeh134. Epub 2004 Apr 30. PMID 15121722
- [Background] Pirotte T, Veyckemans F. Ultrasound-guided subclavian vein cannulation in infants and children: a novel approach. Br J Anaesth. 2007 Apr;98(4):509-14. doi: 10.1093/bja/aem041. Epub 2007 Mar 1. PMID 17332002
- [Background] Iwashima S, Ishikawa T, Ohzeki T. Ultrasound-guided versus landmark-guided femoral vein access in pediatric cardiac catheterization. Pediatr Cardiol. 2008 Mar;29(2):339-42. doi: 10.1007/s00246-007-9066-2. Epub 2007 Sep 13. PMID 17851631
- [Background] Stenzel JP, Green TP, Fuhrman BP, Carlson PE, Marchessault RP. Percutaneous central venous catheterization in a pediatric intensive care unit: a survival analysis of complications. Crit Care Med. 1989 Oct;17(10):984-8. doi: 10.1097/00003246-198910000-00003. PMID 2791583
- [Background] Diggle PJ, Liang KY, Zeger S: Analysis of Longitudinal Data. New York, NY, Oxford University Press, 1995, pp 162-168, 185- 189
- [Background] Johnson EM, Saltzman DA, Suh G, Dahms RA, Leonard AS. Complications and risks of central venous catheter placement in children. Surgery. 1998 Nov;124(5):911-6. PMID 9823406
- [Background] Mansfield PF, Hohn DC, Fornage BD, Gregurich MA, Ota DM. Complications and failures of subclavian-vein catheterization. N Engl J Med. 1994 Dec 29;331(26):1735-8. doi: 10.1056/NEJM199412293312602. PMID 7984193
- [Background] Milling T, Holden C, Melniker L, Briggs WM, Birkhahn R, Gaeta T. Randomized controlled trial of single-operator vs. two-operator ultrasound guidance for internal jugular central venous cannulation. Acad Emerg Med. 2006 Mar;13(3):245-7. doi: 10.1197/j.aem.2005.09.004. Epub 2006 Feb 22. PMID 16495416

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 - Traditional Anatomic Landmark- LM: traditional anatomic landmark CVC placement utilizing palpation and the Seldinger technique
- Group 2 - Ultra Sound US: ultra sound assisted CVC placement
Period: Overall Study
Arm/Group | Group 1 - Traditional Anatomic Landmark- LM | Group 2 - Ultra Sound US
Started | 93 | 119
Completed | 93 | 119
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Two hundred twelve CVC placements were performed and evaluated: 93 during the LM phase and 119 in the US phase.
Groups:
- Group 1 - LM: traditional anatomic landmark CVC placement utilizing palpation and the Seldinger technique
- Group 2 - US: ultra sound assisted CVC placement
- Total: Total of all reporting groups
Arm/Group | Group 1 - LM | Group 2 - US | Total
Number analyzed (Participants) | 93 | 119 | 212
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 93 | 119 | 212
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — Number of patients for whom gender was recorded.
  Participants
    Patients for whom gender was recorded | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Central Line Placement Success
Description: Success was defined as central venous catheter being able to thread into the vessel over the guide wire.
Time Frame: immediate
Population: Population consisted of critically ill children requiring placement of a central venous catheter.
Measure: Number; unit: participants
Arm/Group | Group 1 - LM | Group 2 - US
Number analyzed (Participants) | 93 | 119
participants | 82 | 108
Statistical Analysis 1: Comparison: Group 1 - LM vs Group 2 - US; Test type: Superiority or Other; p < 0.001, Fisher Exact

2. Secondary Outcome: Time to Successful Central Line Placement
Description: Time, in seconds, till successful guide wire placement was achieved.
Time Frame: immediate
Population: Critically ill children requiring central venous access.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Group 1 - LM | Group 2 - US
Number analyzed (Participants) | 93 | 119
seconds | 269 [75 to 900] | 150 [76.5 to 435]

ADVERSE EVENTS:
Groups:
- Group 1 - LM: traditional anatomic landmark central line placement utilizing palpation and the Seldinger technique.
  18/93 (19.4%) had arterial puncture. None was considered serious.
- Group 2 - US: ultra sound assisted central line placement 10/118 (8.5%) had arterial puncture. None was considered serious.
Arm/Group | Group 1 - LM | Group 2 - US
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/119
Other Adverse Events (participants affected / at risk) | 18/93 | 10/119
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - LM (N=93) | Group 2 - US (N=119)
arterial puncture (Blood and lymphatic system disorders) | 18 (18) | 10 (10)

LIMITATIONS AND CAVEATS:
Small sample size. Personnel were aware they were being timed which can bias study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes